CLINICAL TRIAL: NCT07351097
Title: Effect of Adding Mini-squat Exercises at Different Angles to Leg Press Exercise on Quadriceps and Hamstring Strength and H:Q Ratio in Athletes
Brief Title: Adding Mini-squat Exercises to Leg Press Exercise on Quadriceps and Hamstring Strength and H:Q Ratio in Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nasr Awad Abdelkader Othman, Prof, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P.T.REC/012/006017
Record Dates: First submitted 2025-12-31; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (mini-squat at 30° knee flexion and leg press) (Experimental): Fifteen participants will receive mini-squat exercises at 30° knee flexion and leg press exercises
  Interventions: Procedure: mini-squat exercises at 30°
- Group B (mini-squat at 45° knee flexion and leg press) (Active Comparator): Fifteen participants will receive mini-squat exercises at 45° knee flexion and leg press exercises
  Interventions: Procedure: mini-squat exercises at 45°
- Group C (mini-squat at 60° knee flexion and leg press) (Active Comparator): Fifteen participants will receive mini-squat exercises at 60°and leg press exercises
  Interventions: Procedure: mini-squat exercises at 60°
- Group D (Control group: leg press exercise program only) (Placebo Comparator): Fifteen participants will receive leg press exercise program only.
  Interventions: Procedure: leg press exercise

INTERVENTIONS:
Procedure: mini-squat exercises at 30° — mini-squat exercises at 30° knee flexion and leg press exercises
  Arms: Group A (mini-squat at 30° knee flexion and leg press)
Procedure: mini-squat exercises at 45° — mini-squat exercises at 45° knee flexion and leg press exercises
  Arms: Group B (mini-squat at 45° knee flexion and leg press)
Procedure: mini-squat exercises at 60° — mini-squat exercises at 60°and leg press exercises
  Arms: Group C (mini-squat at 60° knee flexion and leg press)
Procedure: leg press exercise — leg press exercise program only
  Arms: Group D (Control group: leg press exercise program only)

SUMMARY:
This study will try to answer the following question:

Will adding mini-squat exercises at different angles (30°,45°, and 60°) to leg press exercise influence quadriceps and hamstring strength and H:Q angle in football players?

DETAILED DESCRIPTION:
Recent studies have highlighted the importance of exercise selection and angle specificity in resistance training, showing that different knee angles result in varied activation patterns in the quadriceps and hamstrings. However, current literature offers limited insight into the effects of integrating mini squat exercises with leg press training on injury prevention and functional outcomes in athletic populations. In particular, there is a lack of literature on how such a combined leg press and mini squat exercise at different angles influences the H:Q ratio, lower limb neuromuscular control, and performance in young male football players. Therefore, the present study aims to examine whether incorporating mini squats performed at varying knee flexion angles into a leg press training program can improve muscle balance and lower limb strength in football players. The findings may provide valuable guidance for physiotherapists, coaches, and sports scientists in developing evidence-based, angle-specific exercise protocols tailored to the functional demands of athletes.

ELIGIBILITY:
Inclusion Criteria:

1. Male football players aged between 18-30 years (Scoz et al., 2021).
2. Body Mass Index (BMI) between 18.5 and 24.9 kg/m² (Walsh et al., 2018 & Sattar& Lean, 2009).
3. Currently training or playing with a registered football club/team.
4. Hamstring-to-Quadriceps (HQ) strength ratio of ≥ 0.6 (Çelebi et al., 2018).
5. Having no oral or injectable non-steroidal anti-inflammatory drugs (NSAID), 2weeks before starting study.
6. Having no oral injectable corticosteroids 3 months before starting the study.

Exclusion Criteria:

1. History of acute or chronic injury to the knee, hip, or ankle joint
2. Undergoing any other rehabilitation or physical therapy programs during the six weeks before starting the study
3. Diagnosed with neurological or systemic disorders affecting muscle function or balance
4. Participation in competitive sports or high-intensity training outside the study protocol during the study period
5. Presence of any contraindication to exercise, such as uncontrolled hypertension or heart conditions.
6. Clinically free from lower limb injuries.
7. Having no history of neurological, cardiovascular, or musculoskeletal disorders.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male football players aged between 18-30 years
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of quadriceps strength | 1.5 months
  * The participant will be seated on the isokinetic dynamometer chair, with proper posture and alignment ensured.
  * The lateral femoral epicondyle (the anatomical axis of the knee joint) will be aligned with the mechanical axis of the dynamometer arm.
  * The lever arm of the dynamometer will be securely attached to the participant's lower leg, just above the ankle, using a padded cuff.
  * The participant will be instructed to perform maximal knee extension against the resistance of the device, moving from a flexed to an extended position.
  * The test will be conducted unilaterally, assessing one leg at a time.
  * The participant will be encouraged to exert maximal effort during each repetition.
  * The isokinetic device will record key outcome measures including peak torque (Nm), average power, and total work for each repetition. These values will be used to quantify quadriceps strength.
Measurement of hamstrings muscle strength | 1.5 months
  All previously described quadriceps muscle evaluation procedures will be applied for the hamstrings muscle strength test; however, the range of motion will be set from full knee extension, and the participant will be instructed to actively bend the knee against the resistance of the device to 90°
Hamstring to quadriceps H:Q ratio calculation | 1.5 months
  The H-Q ratio refers to the relative strength of the hamstring muscles compared to the quadriceps, typically measured under isokinetic conditions (at the same angular velocity). It is calculated as the maximal concentric knee flexion strength divided by maximal concentric knee extension strength.

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Dr.Nasr Abdelkader, Principal Investigator — Cairo Univesity
Locations (1):
- Jazan University Hospital, Jizan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT07351097/Prot_SAP_ICF_000.pdf